CLINICAL TRIAL: NCT02369081
Title: Optimum Treatment for Drug-Resistant Hypertension
Acronym: PATHWAY2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cambridge (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Morris Brown, Professor, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UKCRN 4500; 2008-007149-30 (EudraCT Number)
Record Dates: First submitted 2013-06-11; First posted 2015-02-23 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Hypertension
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Hypertension | interventions — Spironolactone; Bisoprolol; Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Spironolactone (Active Comparator): Each patient will patients will receive in random order 12 weeks treatment with each of the three active drugs (spironolactone, bisoprolol, doxazosin) or placebo. The dose will be doubled at the six week visit half-way through each phase.
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Each patient will patients will receive in random order 12 weeks treatment with each of the three active drugs (spironolactone, bisoprolol, doxazosin) or placebo. The dose will be doubled at the six week visit half-way through each phase
  Interventions: Drug: Placebo
- Doxazosin (Active Comparator): Each patient will patients will receive in random order 12 weeks treatment with each of the three active drugs (spironolactone, bisoprolol, doxazosin) or placebo. The dose will be doubled at the six week visit half-way through each phase
  Interventions: Drug: Doxazosin
- Bisoprolol (Active Comparator): Each patient will patients will receive in random order 12 weeks treatment with each of the three active drugs (spironolactone, bisoprolol, doxazosin) or placebo. The dose will be doubled at the six week visit half-way through each phase
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Spironolactone — Spironolactone 25mg tablet orally once daily for 6 weeks, followed by Spironolactone 50mg tablet orally once daily for a further 6 weeks.
  Arms: Spironolactone
Drug: Bisoprolol — Bisoprolol 5mg tablet orally once each day for 6 weeks, followed by Bisoprolol 10mg tablet orally once each day for a further 6 weeks.
  Arms: Bisoprolol
Drug: Doxazosin — Doxazosin 4mg tablet orally once daily for 6 weeks, followed by Doxazosin 8mg tablet orally once daily for a further 6 weeks.
  Arms: Doxazosin
Drug: Placebo — Placebo treatment for 12 weeks.
  Arms: Placebo

SUMMARY:
This study was recommended by NICE, as part of its 2006 guidance for the treatment of hypertension, and is urgently required to provide evidence for the treatment recommendations in patients with resistant hypertension. The study will be a randomised placebo-controlled double-blind crossover comparison of an α-blocker (α), β-blocker (β), and K+-sparing diuretic (∆).

Patients will have a BP at entry above target on ABPM or home monitoring despite supervised administration of maximum tolerated doses of A+C+D. Over 48 weeks they will then receive, in random order either placebo or two doses each of doxazosin (α), bisoprolol (β) or spironolactone (∆). Each treatment cycle will last 12 weeks, with a forced dose-doubling at 6 weeks.

The time course for the study will be similar to study one. 340 patients will provide 90% power, at α=0.01 to detect a 3 mmHg overall difference in home sBP between any one drug and placebo, with spironolactone hypothesized to be best overall. The study will be able to detect a 6 mmHg difference in sBP between each subject's best and second-best drug predicted by tertile of plasma renin, justifying routine use of the measurement in patients with resistant hypertension.

DETAILED DESCRIPTION:
In published surveys throughout the world the majority of patients with hypertension do not achieve target blood pressure. According to most guidelines including NICE, target blood pressure is 130/80 mmHg in patients with diabetes, 140/90 mmHg in other patients. In the UK there are currently at least 3 million people with treated hypertension whose blood pressure is not controlled. A significant number of these patients will have drug resistant hypertension, defined as:

"a blood pressure that is not adequately controlled to recommended treatment targets despite treatment with maximal recommended and tolerated doses of 3 drugs according to the current BHS/NICE guidelines and treatment algorithm, i.e. (*ACE-inhibitor or *ARB or direct renin inhibitor + *CCB + Diuretic (any diuretic except spironolactone), i.e. A+C+D)".

(*where ACE-inhibitor=angiotensin converting enzyme inhibitor, ARB=angiotensin receptor blocker, CCB=calcium channel blocker)

The causes of treatment resistance are unknown, and the choice of fourth-line drug almost entirely empirical. At present there is little comparative data for available drugs. There is considerable evidence pointing to Na+ retention as a common culprit, and some data supporting additional diuretics, or alpha blockade in resistant hypertension, though mainly added to two rather than three drugs.20,29,30 A retrospective analysis of two-drug combinations in trials reported that it makes no difference what is combined with what. 31 However, this conclusion conflicts with the view that drugs for hypertension fall into two main categories, acting respectively on the renin and volume components of hypertension, and that most benefit can be derived from combining drugs from different categories.10,32

Despite the successful adoption of the BHS/NICE treatment algorithm for the treatment of hypertension, there remains substantial clinical uncertainty about the preferred clinical management of people with drug resistant hypertension. This is an important question because such patients are at the highest risk for cardiovascular events. The current guidelines acknowledge that there is currently no adequate clinical trial evidence upon which to base recommendations for the preferred 4th line drug treatment for those with resistant hypertension.

It is possible that it makes no difference what drug is added as fourth-line treatment and that the response, on average, will be the same for all classes. Alternatively, it is also possible that one class of drug will always be superior to all the others because the mechanism underpinning resistant hypertension is common to all patients. In this regard, a popular view is that resistant hypertension is invariably due to excessive sodium retention and thus "further diuretic therapy" will always be the most effective treatment. A third possibility is that resistant hypertension is a heterogeneous state and that the study of average responses in cohorts in clinical studies masks substantial individual patient differences.

With regard to this, this study will address the hypothesis that the renin status of the patient defines the response to 4th line treatment in resistant hypertension, i.e. that low renin predicts sodium retention and the best response to diuretic therapy, whereas high renin predicts a better response to drugs that suppress renin, i.e. a β-blocker.

Hypothesis and Novel Aspects of the Trial

The primary hypothesis of the study is that the commonest cause of resistant hypertension is excessive Na+-retention, and that further diuretic therapy (spironolactone used in this study) will be superior to other potential "add-on drugs" for people with inadequate blood pressure control despite treatment with optimal or highest tolerated doses of the three drug classes recommended by the BHS/NICE treatment algorithm, i.e. A+C+D.

The main secondary objective is to use plasma renin measurements to evaluate an 'α, β, ∆' rule for the selection of the 4th line drug for patients with drug resistant hypertension - where α represents α-blockade, β represents β-blockade and ∆ represents "further diuretic therapy" as cited above. The main secondary hypothesis states that plasma renin (measured on a background of 3 drugs, i.e. A+C+D), will predict the most effective 4th line drug. We propose that:

α-blockade will be the most effective 4th line drug at lowering BP in patients in the mid-tertile of plasma renin, expected to be ≥20mU/L but <100mU/L; β-blockade will be the most effective drug when renin is in the top tertile (expected to be ≥100Mu/L) as the drug blocks renin secretion; Further diuretic therapy with spironolactone will be most effective when plasma renin is in the lowest tertile (expected to be <20mU/L), indicative of excessive sodium retention.

The study will also evaluate whether the routine use of plasma renin to predict best treatment in individual patients with resistant hypertension will be more cost-effective than using further diuretic therapy indiscriminately as the preferred 4th line drug for all patients.

Finally the study will investigate whether non-invasive assessment of haemodynamic parameters indicative of sodium retention and volume status, i.e. cardiac output, peripheral resistance and bioimpedance, can be used to predict the response to each drug in the α, β, ∆ sequence.

ELIGIBILITY:
Patients must meet ALL inclusion criteria

* M/F 18-79 years
* Patients with hypertension not controlled to target: clinic systolic BP ≥ 5 mmHg above target (i.e. ≥ 140 mmHg for non-diabetic hypertensives or ≥ 135 mmHg for diabetics), under one of the following conditions:

  1. Treatment for at least 3 months with lisinopril 20 mg (A) + amlodipine 10 mg (C) + bendroflumethiazide 2.5 mg (D) or their equivalents
  2. Patients who have received the three drugs or equivalents specified in a), and are either intolerant to one category, or tolerate only a lower dose (e.g. amlodipine 5 mg or lisinopril 10 mg)
  3. Patients receiving the three drugs or equivalents specified in a), who are receiving additional drugs for their hypertension, may be included if the investigator: 1) feels it is appropriate to stop these additional drugs at the screening visit and 2) anticipates that the BP criteria for inclusion will be met when re-checked at the baseline visit Patients may be included if the PI anticipates BP criteria for inclusion will be met at randomisation.
* Patients with a home systolic BP average of >130 mmHg or within 15mmHg of clinic BP over the 4 days prior to the baseline visit.

Exclusion;

* Inability to give informed consent;
* Participation in a clinical study involving an investigational drug or device within 4 weeks of screening;
* Secondary or accelerated hypertension;
* Type 1 diabetes;
* eGFR<45 mls/min;
* Plasma potassium outside of normal range on two successive measurements during screening;
* Pregnancy, planning to conceive, or women of child-bearing potential not taking adequate contraception
* Anticipated change of medical status during the trial - Absolute contra-indication to study drugs or previous intolerance of trial therapy;
* Sustained atrial fibrillation;
* Recent cardiovascular event requiring hospitalisation
* Suspected non-adherence to antihypertensive treatment
* Requirement for study drug for reason other than to treat hypertension, - Current therapy for cancer;
* Concurrent chronic illness, likely to preclude 52 week participation in the study;
* Clinic Systolic BP >200 mmHg or diastolic BP >120mmHg, with PI discretion to override if home BP measurements are lower
* Any concomitant condition that may adversely affect the safety/ efficacy of study drug or severely limit that patients life-span or ability to complete the study
* Treatment with any of the following medications;

  1. Oral corticosteroids within 3 months of screening. Treatment with systemic corticosteroids is also prohibited during study participation;
  2. Chronic stable use, or unstable use of NSAIDs (other than low dose aspirin) is prohibited. Chronic use defined as >3 consecutive or non-consecutive days of treatment per week. In addition intermittent use of NSAIDs is strongly discouraged; if required, must not be used for more than a total of 2 days. For those requiring analgesics; paracetamol is recommended.
  3. The use of short acting nitrates is permitted, but must not be taken within 4 hours of screening or subsequent visits
  4. The use of long acting nitrates is permitted but dose must be stable for at least 2 weeks prior to screening and randomisation;
  5. The use of sympathomimetic decongestants is permitted;but not within 1 day prior to any study visit/BP assessment;
  6. The use of theophylline is permitted but dose must be stable for 4 weeks prior to screening and throughout the study;
  7. The use of phosphodiesterase type V inhibitors is permitted; however study participants must refrain from taking these medications for at least 1 day prior to screening or any subsequent study visits;
  8. The use of alpha-blockers is not permitted, with the exception of afluzosin and tamsulosin for prostatic symptoms
* A pill count will be made at the end of the 4 week run-in period and those with adherence <70% will be excluded from randomisation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2009-05; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Treatment arm comparison according to home blood pressure measurement | 48 weeks
  We will adopt a hierarchical procedure to test, in order, the differences in home systolic BP between spironolactone and
  1. placebo
  2. the average of the other two active drugs
  3. each of the other two drugs. The second and third tests will be carried out if and only if the preceding test(s) are significant (P<0.05).
  We shall use a mixed model to analyse home BP, with unstructured covariances for the repeated measures across the two doses for each treatment within a patient. The model will include terms for gender, age, height, weight, smoking history and a diagnosis of diabetes at baseline. We will also adjust for baseline BP.

SECONDARY OUTCOMES:
Measurement of plasma renin as predictor of effective treatment | 48 weeks
  The difference in home systolic BP averages between the best drug predicted by the patient's plasma renin (according to the 'α, β, ∆' rule cited above) and further diuretic therapy;ie with spironolactone, which we have predicted will be the most effective treatment on average.

OTHER OUTCOMES:
Cardiac Index (L/min/m2) measured at baseline and the end of the 4 treatment cycles | 48 weeks
  This is assessed non-invasively. We hypothesize that patients in the highest quartile of cardiac index at baseline will respond more to beta-blockade (bisoprolol) than to other treatments, and that this parameter will be reduced more by beta-blockade than by other treatments.
Systemic Vascular Resistance Index (dyne/sec/cm-5) measured at baseline and the end of the 4 treatment cycles | 48 weeks
  This is assessed non-invasively. We hypothesize that patients in the highest quartile of systemic vascular resistance at baseline will respond more to alpha-blockade (doxazosin) than to other treatments, and that this parameter will be reduced more by alpha-blockade than by other treatments.
Thoracic fluid content (KOhm-1) measured at baseline and the end of the 4 treatment cycles | 48
  This is assessed non-invasively. We hypothesize that patients in the highest quartile of thoracic fluid content at baseline will respond more to additional diuretic (spironolactone) than to other treatments, and that this parameter will be reduced more by spironolactone than by other treatments.
Pulse wave velocity (m/s) measured at baseline and the end of the 4 treatment cycles | 48
  We hypothesize that this parameter will be reduced more by spironolactone than by other treatments.
Supine central systolic pressure (mmHg) measured at baseline and the end of the 4 treatment cycles | 48
  We hypothesize that this parameter will be reduced more by spironolactone than by other treatments.
Augmentation index (%) measured at baseline and the end of the 4 treatment cycles | 48
  We hypothesize that this parameter will be reduced more by spironolactone than by other treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Prof MJ Brown, Principal Investigator — University of Cambridge
Locations (16):
- United Kingdom (16):
  - NHS Ayrshire, Ayrshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University of Birmingham, Birmingham
  - University of Cambridge - Addenbrookes Hospital, Cambridge
  - NHS Tayside/University of Dundee, Dundee
  - NHS Lothian/University of Edinburgh, Edinburgh
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - NHS Greater Glasgow and Clyde/University of Glasgow, Glasgow
  - Ixworth GP Practice, Ixworth
  - University Hospitals of Leicester NHS Trust, Leicester
  - Barts and the London School of Medicine and Dentistry, London
  - Guys and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Norfolk and Norwich University Hospital NHS Trust, Norwich
  - West Hertfordshire Hospitals NHS Trust, Watford

REFERENCES:
- [Background] NICE/BHS. CG34 Hypertension - NICE guideline (all the recommendations). http://www.nice.org.uk/guidance/CG34/niceguidance /pdf/english 2006
- [Background] Dickerson JE, Hingorani AD, Ashby MJ, Palmer CR, Brown MJ. Optimisation of antihypertensive treatment by crossover rotation of four major classes. Lancet. 1999 Jun 12;353(9169):2008-13. doi: 10.1016/s0140-6736(98)07614-4. PMID 10376615
- [Background] Deary AJ, Schumann AL, Murfet H, Haydock SF, Foo RS, Brown MJ. Double-blind, placebo-controlled crossover comparison of five classes of antihypertensive drugs. J Hypertens. 2002 Apr;20(4):771-7. doi: 10.1097/00004872-200204000-00037. PMID 11910315
- [Background] Taler SJ, Textor SC, Augustine JE. Resistant hypertension: comparing hemodynamic management to specialist care. Hypertension. 2002 May;39(5):982-8. doi: 10.1161/01.hyp.0000016176.16042.2f. PMID 12019280
- [Background] Kaplan NM. Resistant hypertension. J Hypertens. 2005 Aug;23(8):1441-4. doi: 10.1097/01.hjh.0000174968.72212.ac. PMID 16003165
- [Background] Black HR, Keck M, Meredith P, Bullen K, Quinn S, Koren A. Controlled-release doxazosin as combination therapy in hypertension: the GATES study. J Clin Hypertens (Greenwich). 2006 Mar;8(3):159-66; quiz 167-8. doi: 10.1111/j.1524-6175.2006.04811.x. PMID 16522992
- [Background] Law MR, Wald NJ, Morris JK, Jordan RE. Value of low dose combination treatment with blood pressure lowering drugs: analysis of 354 randomised trials. BMJ. 2003 Jun 28;326(7404):1427. doi: 10.1136/bmj.326.7404.1427. PMID 12829555
- [Background] Brown MJ, Cruickshank JK, Dominiczak AF, MacGregor GA, Poulter NR, Russell GI, Thom S, Williams B; Executive Committee, British Hypertension Society. Better blood pressure control: how to combine drugs. J Hum Hypertens. 2003 Feb;17(2):81-6. doi: 10.1038/sj.jhh.1001511. PMID 12574784
- [Derived] Williams B, MacDonald TM, Morant SV, Webb DJ, Sever P, McInnes GT, Ford I, Cruickshank JK, Caulfield MJ, Padmanabhan S, Mackenzie IS, Salsbury J, Brown MJ; British Hypertension Society programme of Prevention And Treatment of Hypertension With Algorithm based Therapy (PATHWAY) Study Group. Endocrine and haemodynamic changes in resistant hypertension, and blood pressure responses to spironolactone or amiloride: the PATHWAY-2 mechanisms substudies. Lancet Diabetes Endocrinol. 2018 Jun;6(6):464-475. doi: 10.1016/S2213-8587(18)30071-8. Epub 2018 Apr 11. PMID 29655877
- [Derived] Williams B, MacDonald TM, Morant S, Webb DJ, Sever P, McInnes G, Ford I, Cruickshank JK, Caulfield MJ, Salsbury J, Mackenzie I, Padmanabhan S, Brown MJ; British Hypertension Society's PATHWAY Studies Group. Spironolactone versus placebo, bisoprolol, and doxazosin to determine the optimal treatment for drug-resistant hypertension (PATHWAY-2): a randomised, double-blind, crossover trial. Lancet. 2015 Nov 21;386(10008):2059-2068. doi: 10.1016/S0140-6736(15)00257-3. Epub 2015 Sep 20. PMID 26414968
- [Derived] Williams B, MacDonald TM, Caulfield M, Cruickshank JK, McInnes G, Sever P, Webb DJ, Salsbury J, Morant S, Ford I, Brown MJ. Prevention And Treatment of Hypertension With Algorithm-based therapy (PATHWAY) number 2: protocol for a randomised crossover trial to determine optimal treatment for drug-resistant hypertension. BMJ Open. 2015 Aug 7;5(8):e008951. doi: 10.1136/bmjopen-2015-008951. PMID 26253568